CLINICAL TRIAL: NCT05105529
Title: Pulmonary and Vascular Adaptations to a 5-days Exercise Protocol in Ozone in Physically Active Individuals With Asthma and Exercise-induced Bronchoconstriction
Brief Title: Adaptation to Ozone in Individuals With Asthma/Exercise-induced Bronchoconstriction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Koehle, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H21-01183
Record Dates: First submitted 2021-09-28; First posted 2021-11-03 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Asthma; Asthma, Exercise-Induced; Exercise Induced Asthma; Exercise Induced Bronchospasm
Keywords: Ozone; Air pollution; Asthma; Exercise-induced bronchoconstriction
MeSH Terms: conditions — Asthma; Asthma, Exercise-Induced | interventions — Exercise; Ozone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Air quality condition (Ozone and filtered air) will be double-blinded; Participants will not be told at any time before the study completion to which group they are assigned (intervention or sham)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone (O3) group (Experimental): Participants of the experimental group will perform sub-maximal exercise (60% of VO2max for 30 minutes) on a cycle ergometer while inhaling 170ppb ozone delivered continuously during each exercise session.
  Interventions: Behavioral: Exercise; Other: Ozone
- Filtered Air (Sham Comparator): Participants of the sham group will also perform sub-maximal exercise (60% of VO2max for 30 minutes) on a cycle ergometer similar to intervention. However, only in this group, the ozone generator will not be activated so that just filtered air will be delivered to the participant while performing each exercise session.
  Interventions: Behavioral: Exercise; Other: Filtere Air

INTERVENTIONS:
Behavioral: Exercise — Cycling at 60% of VO2max on a cycle ergometer for 30 minutes
Other: Ozone — Breathing 170ppb ozone
  Arms: Ozone (O3) group
Other: Filtere Air — Breathing filtered air
  Arms: Filtered Air

SUMMARY:
Researchers found that impairments in the cardiopulmonary system caused by acute exposure to ozone were outweighed by repeated exposures to ozone. The goal of this study is to confirm there will be an adaptation similar to what was previously proved but in individuals with asthma and exercise-induced bronchoconstriction (EIB). The purpose is to examine adaptive responses in a randomized cross-over trial in which physically active individuals will perform submaximal exercise on five days in ozone and filtered air exposures separated by a washout period.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active individuals
* Diagnosed asthma and/or mild exercise-induced bronchoconstriction: defined by an FEV1 fall equal to or greater than 10% but lower than 25% in the eucapnic hyperventilatory test.
* Able to securely perform a maximal exercise test (responded 'no' to all questions on the PAR-Q+ questionnaire)
* Able to communicate in English

Exclusion Criteria:

* Diagnosed with any cardiorespiratory or vascular diseases
* Pregnant or potentially pregnant
* Non-smoking
* Lower limb musculoskeletal injury or lower limb limitation to cycle on a bicycle ergometer
* Recent respiratory symptoms or upper tract infection within 4 weeks
* On vitamin (e.g., C or E) supplementation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in FEV1 from baseline to 10 minutes after exercise | Measured at baseline and 10 minutes after each exercise bout
  Measurement of pulmonary function: forced exhaled volume in the first second (FEV1) in liters
Change in FVC from baseline to 10 minutes after exercise | Measured at baseline and 10 minutes after each exercise bout
  Measurement of pulmonary function: forced vital capacity (FVC) in liters
Change in FEF25-75 from baseline to 10 minutes after exercise | Measured at baseline and 10 minutes after each exercise bout
  Measurement of pulmonary function: forced expiratory flow at 25-75% of pulmonary volume in liters per second (L/s)

SECONDARY OUTCOMES:
Change in Pulse Wave Velocity (PWV) from baseline to 20 minutes after exercise | Measured at baseline and 20 minutes after each exercise bout
  Velocity (in meters per second) at which the blood pressure pulse propagates through set points in the circulatory system
Change in Fraction of exhaled nitric oxide (FeNO) from baseline to 5 minutes after exercise | Measured at baseline and 5 minutes after each exercise bout
  Non-invasive airway inflammation biomarker (in part per billion, ppb)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koehle, MD PhD, Principal Investigator — Professor
Locations (2):
- Canada (2):
  - Environmental Physiology Laboratory, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No